CLINICAL TRIAL: NCT00399074
Title: Presumptive Treatment With Sulfadoxine- Pyrimethamine Versus Weekly Chloroquine for Malaria Prophylaxis in Children With Sickle Cell Anemia
Brief Title: Sulfadoxine- Pyrimethamine Versus Weekly Chloroquine for Malaria Prevention in Children With Sickle Cell Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: James K Tumwine, Department of Paediatrics and Child Health Makerere University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2004/HD11/1353U
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Sickle Cell Anemia; Malaria
Keywords: Sickle Cell anemia; Malaria; Presumptive treatment; Sulfadoxine- pyrimethamine; Children; Uganda
MeSH Terms: conditions — Anemia, Sickle Cell; Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- chloroquine (No Intervention): Weekly CQ
- Sulfadoxine-pyrimethamine (No Intervention): Monthly SP
  Interventions: Drug: sulfadoxine pyrimethamine

INTERVENTIONS:
Drug: sulfadoxine pyrimethamine — Monthly SP
  Other Names: SP
  Arms: Sulfadoxine-pyrimethamine

SUMMARY:
Malaria is fatal and increases the risk of death among children with sickle cell anemia. Chemoprophylaxis significantly improves quality of life in these children. In Uganda Chloroquine is the drug of choice for prophylaxis and yet it's effectiveness is limited due to high levels of resistance throughout the country. Intermittent presumptive treatment with sulfadoxine - Pyrimethamine a new approach to malaria prevention, has shown great potential in reducing incidence of malaria and anaemia among high risk groups such as pregnant women and infants. However no studies have been done in Uganda to determine if presumptive treatment with sulfadoxine- pyrimethamine reduces the incidence of malaria in children with sickle cell anaemia.

Hypothesis : Presumptive treatment with sulfadoxine- Pyrimethamine is better than weekly chloroquine in reducing incidence of malaria in children with sickle cell anaemia.

DETAILED DESCRIPTION:
Malaria is fatal and increases the risk of death among children with sickle cell anemia. Chemoprophylaxis significantly improves quality of life in these children. In Uganda Chloroquine is the drug of choice for prophylaxis and yet it's effectiveness is limited due to high levels of resistance throughout the country. Intermittent presumptive treatment with sulfadoxine - pyrimethamine a new approach to malaria prevention, has shown great potential in reducing incidence of malaria and anemia among high risk groups such as pregnant women and infants. However no studies have been done in Uganda to determine if presumptive treatment with sulfadoxine- pyrimethamine reduces incidence of malaria among high risk group such as children with sickle cell anaemia.

We calculated a sample size of 110 patients in each group for a power of 95% assuming that the incidence of malaria in children receiving weekly chloroquine will be 0.36 and those receiving presumptive treatment with sulfadoxine - pyrimethamine the incidence would be 0.16 according to (schellenberg et al )

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 12 years attending sickle cell clinic in Mulago Hospital during the study period with a negative peripheral smear for parasites, adherence to appointment visits, consent by care takers to participate in the study.

Exclusion Criteria:

* Patients with known allergy to sulfonamides, Patients with severe illnesses requiring urgent admission, Patients with documented treatment for malaria in the past one month with Sulfadoxine- Pyrimethamine. Patients on cotrimoxazole prophylaxis

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Malaria episodes | 4 weeks

SECONDARY OUTCOMES:
Malaria related admissions | 1 month
Adverse drug effects | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Nakibuuka, MBChB, Principal Investigator — Department of Paediatrics and Child Health , Makerere University; Grace Ndeezi, M.Med, Principal Investigator — Department of Paediatrics and Child Health, Makerere University; Deborah Nakiboneka, M.Med, Principal Investigator — Department of Paediatrics and Child Health, Makerere University; Christopher Ndugwa, PhD, Principal Investigator — Department of paediatrics and Child Health, Makerere University; James Tumwine, PhD, Principal Investigator — Department of Paediatrics and Child Health, Makerere University
Locations (1):
- Mulago Hospital, Kampala, Central Region, Uganda

REFERENCES:
- [Background] Schellenberg D, Menendez C, Kahigwa E, Aponte J, Vidal J, Tanner M, Mshinda H, Alonso P. Intermittent treatment for malaria and anaemia control at time of routine vaccinations in Tanzanian infants: a randomised, placebo-controlled trial. Lancet. 2001 May 12;357(9267):1471-7. doi: 10.1016/S0140-6736(00)04643-2. PMID 11377597
- [Background] Massaga JJ, Kitua AY, Lemnge MM, Akida JA, Malle LN, Ronn AM, Theander TG, Bygbjerg IC. Effect of intermittent treatment with amodiaquine on anaemia and malarial fevers in infants in Tanzania: a randomised placebo-controlled trial. Lancet. 2003 May 31;361(9372):1853-60. doi: 10.1016/s0140-6736(03)13504-0. PMID 12788572
- [Background] Cisse B, Sokhna C, Boulanger D, Milet J, Ba el H, Richardson K, Hallett R, Sutherland C, Simondon K, Simondon F, Alexander N, Gaye O, Targett G, Lines J, Greenwood B, Trape JF. Seasonal intermittent preventive treatment with artesunate and sulfadoxine-pyrimethamine for prevention of malaria in Senegalese children: a randomised, placebo-controlled, double-blind trial. Lancet. 2006 Feb 25;367(9511):659-67. doi: 10.1016/S0140-6736(06)68264-0. PMID 16503464